CLINICAL TRIAL: NCT06525987
Title: Telecoached Exercise Intervention for Connectivity Enhancement in Small Vessel Disease (TELECONNECT-SVD): a Randomized Clinical Trial
Brief Title: Telecoached Exercise Intervention for Connectivity Enhancement in Small Vessel Disease (TELECONNECT-SVD)
Acronym: TELECONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Simona Sacco, Full Professor of Neurology, University of L'Aquila
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Not yet determined
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lacunar Stroke; Small Vessel Cerebrovascular Disease
MeSH Terms: conditions — Stroke, Lacunar; Cerebral Small Vessel Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The trial will adopt a "wait list" delish in which one group will be randomized to immediate intervention while the other group will be randomized to delayed intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by investigators blinded to participants' allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): Participants will be allocated to physical activity intervention during the 24 weeks of follow-up.
  Interventions: Behavioral: Physical activity
- Delayed intervention (Other): Participants will not be randomized to physical activity intervention during the first 24 weeks of follow-up. They will be randomized after the 24 weeks of follow-up.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Randomization to a 24-week physical exercise program
  Other Names: Physical activity (delayed)

SUMMARY:
The TELECONNECT-SVD study is a prospective, randomized, multicenter trial aimed at testing the efficacy of a remotely delivered exercise protocol on brain functional connectivity in patients with small vessel disease (SVD)-related ischemic stroke. The study will recruit patients aged ≥60 with a history of lacunar stroke, minimal disability (modified Rankin Scale score 0-1), and low physical activity levels.

The trial will include 60 participants randomized 1:1 to either a 24-week telecoached exercise intervention or usual care. The exercise program consists of multicomponent physical exercises delivered remotely twice a week. Assessments will be conducted at baseline, 12 weeks, 24 weeks, and 48 weeks.

Primary outcomes include changes in brain functional connectivity assessed by high-density EEG and improvements in physical fitness measured by the Senior Fitness Test. Secondary outcomes encompass changes in physical activity levels, anthropometric measurements, and vital signs.

The study employs a "wait list" design, where the control group receives the intervention after the initial 24-week period. This approach allows for assessment of the intervention's immediate effects and the retention of benefits after cessation.

Key features of the protocol include:

* Use of telecoaching to enhance adherence to the exercise program
* Comprehensive assessment of brain connectivity using advanced EEG analysis techniques
* Focus on patients with SVD, who may benefit significantly from exercise interventions
* Evaluation of both neurophysiological and clinical outcomes

The study aims to provide evidence for the potential benefits of exercise in enhancing brain connectivity and physical fitness in SVD patients, potentially informing future treatment guidelines and preventive strategies for this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years;
* History of lacunar stroke occurred between 3 months and 10 years from screening and confirmed by neuroimaging or clinical data by an expert stroke physician;
* Modified Rankin Scale (mRS) score of 0-1, indicating no symptoms or no significant disability;
* A level of physical activity below recommended targets, i.e. <150 minutes per week of moderate-to-vigorous exercise (24);
* Ability to sign informed consent.

Exclusion Criteria:

* Uncontrolled hypertension;
* Heart disease impairing the possibility of safely following an exercise protocol at the discretion of the treating physician;
* Primary or secondary epilepsy;
* Prostheses, implants, and any device that might impair the performance of either high-density electroencephalogram or the exercise intervention;
* Cognitive impairment (Mini Mental State Examination score ≤26 at follow-up);
* Lack of access to Internet-based facilities or poor technological alphabetization impairing the adherence to the trial protocol;
* Any major physical or psychiatric comorbidity that in the judgement of the treating physician might compromise the ability to undergo an exercise intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Senior Fitness Test score | 24 weeks
  Change in the Senior Fitness score from before to after the 24-week physical exercise intervention

SECONDARY OUTCOMES:
Change in International Physical Activity Questionnaire (IPAQ) score | 24 weeks
  Change in International Physical Activity Questionnaire (IPAQ) score from before to after the 24-week physical exercise intervention
Change in Body Mass Index | 24 weeks
  Change in Body Mass Index score from before to after the 24-week physical exercise intervention
Change in blood pressure | 24 weeks
  Change in blood pressure from before to after the 24-week physical exercise intervention
Change in heart rate | 24 weeks
  Change in heart rate from before to after the 24-week physical exercise intervention

OTHER OUTCOMES:
Change in brain functional connectivity | 24 weeks
  Overall brain functional connectivity in the resting state assessed via high-density electroencephalogram

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Neurologia e Stroke Unit, Avezzano, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be available from the central contact person upon reasonable request.